CLINICAL TRIAL: NCT02835989
Title: Community Paramedicine at Home (CP @Home)
Brief Title: Community Paramedicine at Home
Acronym: CP@Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2153
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Cardiovascular Disease; Diabetes Mellitus; Accidental Falls; Social Isolation; Food Insecurity
Keywords: Community Paramedicine; Paramedic; Emergency Medical Services; High Frequency Callers; Lift Assists
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Social Isolation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CP@Home Intervention (Experimental): The experimental group will receive the CP@Home program. The main elements of this program include BP assessment, diabetes risk assessment, falls risk assessment, heart failure risk assessment, neurologic assessment, psychiatric assessment, depression screening, health-related quality of life analysis (including pain, mobility, anxiety/depression, ADLs), social isolation screening, and food and income security. The program is targeted at referrals to appropriate community resources, identification and referral of high-risk patients to their family physician (FP), as well as regular communication of participants' health information to their physician.
  The intervention will be implemented by community paramedics from the local paramedic service who have undergone a structured training program (4 hours of online, interactive training modules, including case studies and the observation of an intervention visits led by another paramedic) to assure intervention fidelity.
  Interventions: Other: CP@Home
- Control (No Intervention): Usual Care

INTERVENTIONS:
Other: CP@Home — Community paramedics (CPs) will be assigned to visiting the participants for a first time the week following the initial EMS call. Participants will complete the informed consent process with a CP on their first visit. This visit will also include a full assessment and risk analysis that will take approximately 90 minutes and will be located in the participant's home. As a result of the initial visit, the CP will make all relevant clinical referrals and decisions based on predetermined @Home algorithms. A second visit will be made to the participant 2-4 weeks following the initial call for a streamlined follow-up and reassessment during a 30 minute period. A final visit will be made 6-8 weeks following the initial call for a final evaluation of their situation. It is anticipated the patient will be discharged from the CP@Home program at this point. If the patient calls EMS following the third visit, if they meet the inclusion criteria, they will be re-entered into the CP@Home program.
  Arms: CP@Home Intervention

SUMMARY:
Community Paramedicine @Home (CP@Home) is a novel community paramedicine health assessment program for high users of Emergency Medical Services (EMS). Individuals who have been identified as active callers to EMS, individuals who have called EMS for lift-assists, and direct paramedic referrals are referred into the community paramedicine home visit program. The program will focus on in-home chronic disease management, community health service connections, and EMS usage education. Aside from chronic disease management, aspects of the program include health-related quality of life, social isolation and other social determinants of health. Participants in the program will have up to 3 one-on-one home visits from a community paramedic to ultimately reduce repeat EMS calls and improve their overall health.

ELIGIBILITY:
Inclusion Criteria:

* 3 or more EMS calls in the last 6 months from intervention start date AND active caller in the last 30 days OR
* Any call for a lift assist to EMS in the past 30 days OR
* Paramedic referral into program (identified by paramedic through usual practice)

Exclusion Criteria:

* Individuals living in long term care facilities
* Individuals currently involved in a home visit or social navigator program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2826 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in number of repeat EMS calls | Baseline and 1 year
  Individual-level change in EMS call rate resulting in ambulance dispatch (pre-post intervention)

SECONDARY OUTCOMES:
Change in number of ED presentations | Baseline and 1 year
  Individual-level change in number of ED presentations (pre-post)
Change in number of hospital admissions | Baseline and 1 year
  Individual-level change in number of hospital admissions (pre-post)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Agarwal, MBBS MRCGP CCFP PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agarwal G, Angeles R, Brar J, Pirrie M, Marzanek F, McLeod B, Thabane L. Effectiveness of the community paramedicine at home (CP@home) program for frequent users of emergency medical services in Ontario: a randomized controlled trial. BMC Health Serv Res. 2024 Nov 25;24(1):1462. doi: 10.1186/s12913-024-11952-7. PMID 39587610
- [Derived] Agarwal G, Pirrie M, McLeod B, Angeles R, Tavares W, Marzanek F, Thabane L. Rationale and methods of an Evaluation of the Effectiveness of the Community Paramedicine at Home (CP@home) program for frequent users of emergency medical services in multiple Ontario regions: a study protocol for a randomized controlled trial. Trials. 2019 Jan 23;20(1):75. doi: 10.1186/s13063-018-3107-4. PMID 30674347